CLINICAL TRIAL: NCT02622191
Title: Segmental Analysis of Retinal Layers and Measurement of Lamina Cribrosa Thickness in Patients With Asymmetric Primary Open-Angle Glaucoma
Brief Title: Analysis of the Eye in Patients With Primary Open-Angle Glaucoma and a Visual Field Defect in One Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-229
Record Dates: First submitted 2015-11-17; First posted 2015-12-04 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Glaucoma
Keywords: Glaucoma; Optical Coherence Tomography; Primary Open Angle Glaucoma; Visual Field
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-angle glaucoma (Experimental): Participants with primary open-angle glaucoma and an abnormal visual field defect in one eye. Spectral domain Optical Coherence Tomography will be obtained from the effected eye and fellow eye of each glaucoma patient.
  Interventions: Device: Spectral domain Optical Coherence Tomography
- Healthy Controls (Experimental): Participants without glaucoma and no other eye diseases. Spectral domain Optical Coherence Tomography will be obtained from eyes of each healthy control.
  Interventions: Device: Spectral domain Optical Coherence Tomography

INTERVENTIONS:
Device: Spectral domain Optical Coherence Tomography — Undilated peripapillary circular optic nerve scans and horizontal and vertical SD-OCT B-scan images centered on the fovea were acquired using Spectralis Heidelberg Retinal Angiography (HRA)+OCT (Heidelberg Engineering GmbH, Heidelberg, Germany).
  Other Names: SD-OCT

SUMMARY:
The study aims to further understand glaucoma pathogenesis and progression by utilizing enhanced depth imaging optical coherence tomography to visualize and measure lamina cribrosa in vivo and segmentation technology to accurately delineate and measure boundaries of the retinal layers. Investigators will elaborate further on key concepts of lamina cribrosa thickness and trans-synaptic degeneration.

DETAILED DESCRIPTION:
Two important areas of the eye that need investigation in order to further understanding of glaucoma. First is the retina (part of the eye that converts images from the eye's optical system into electrical impulses sent along the optic nerve to the brain). Newer technology, Spectral Domain Optical Coherence Tomography (SD-OCT), allows us to look at different layers of the retina and carefully measure thickness of each layer. Second area is lamina cribrosa (a portion of the white part of the eye which has nerve fibers passing through it connecting the eye to the brain). If lamina cribrosa is thin, it is possible it may bend easily and disrupt nerve fibers. SD-OCT allows measurement of lamina cribrosa thickness.

Findings will help monitor changes that occur in the eye as a result of glaucoma.

Individuals with primary open-angle glaucoma and unilateral visual field defects were chosen as the main patient population (in addition to normal controls). By approximating each participants baseline anatomy using the fellow, "internal control" eye, investigators will be able to better determine if any changes occur in the macula or the lamina cribrosa as a result of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Best-corrected visual acuity of 20/40 or better
* No media opacities
* Spherical equivalent refractive errors in a range of -6 to +6 diopters
* Cylinder correction within 3.0 diopters.

Exclusion Criteria:

* Age < 18 years old
* Visual Acuity < 20/40
* Nuclear sclerosis > +2
* Corneal diseases
* Contact lens use
* History of posterior segment intraocular surgery
* Systemic or ocular diseases that can cause visual field loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L J Katz, MD, Principal Investigator — Wills Eye Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zangalli CS, Ahmed OM, Waisbourd M, H Ali M, Cvintal V, Affel E, Gupta L, Katz LJ, C Sergott R. Segmental Analysis of Macular Layers in Patients With Unilateral Primary Open-Angle Glaucoma. J Glaucoma. 2016 Apr;25(4):e401-7. doi: 10.1097/IJG.0000000000000336. PMID 26550975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with unilateral primary open-angle glaucoma (POAG) were recruited from the Glaucoma Service at Wills Eye Hospital, Philadelphia, PA, USA. Healthy controls were recruited from staff, friends and family. All participants were recruited between November 2012 and February 2013.
Groups:
- Open-angle Glaucoma: Participants with primary open-angle glaucoma and an abnormal visual field defect in one eye. Spectral domain Optical Coherence Tomography will be obtained from the effected eye and fellow eye of each glaucoma patient.
  Spectral domain Optical Coherence Tomography (SD-OCT): Undilated peripapillary circular optic nerve scans and horizontal and vertical SD-OCT B-scan images centered on the fovea were acquired using Spectralis Heidelberg Retinal Angiography (HRA)+OCT (Heidelberg Engineering GmbH, Heidelberg, Germany).
- Healthy Controls: Participants without glaucoma and no other eye diseases. Spectral domain Optical Coherence Tomography will be obtained from eyes of each healthy control.
  Spectral domain Optical Coherence Tomography (SD-OCT): Undilated peripapillary circular optic nerve scans and horizontal and vertical SD-OCT B-scan images centered on the fovea were acquired using Spectralis Heidelberg Retinal Angiography (HRA)+OCT (Heidelberg Engineering GmbH, Heidelberg, Germany).
Period: Overall Study
Arm/Group | Open-angle Glaucoma | Healthy Controls
Started | 19 | 14
Completed | 19 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-angle Glaucoma: Participants with primary open-angle glaucoma and an abnormal visual field defect in one eye. Spectral domain Optical Coherence Tomography will be obtained from the effected eye and fellow eye of each glaucoma patient.
  Spectral domain Optical Coherence Tomography: Undilated peripapillary circular optic nerve scans and horizontal and vertical SD-OCT B-scan images centered on the fovea.
- Healthy Controls: Participants without glaucoma and no other eye diseases. Spectral domain Optical Coherence Tomography will be obtained from eyes of each healthy control.
  Spectral domain Optical Coherence Tomography: Undilated peripapillary circular optic nerve scans and horizontal and vertical SD-OCT B-scan images centered on the fovea.
- Total: Total of all reporting groups
Arm/Group | Open-angle Glaucoma | Healthy Controls | Total
Number analyzed (Participants) | 19 | 14 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 13 | 10 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Lamina Cribrosa (Boundaries of the Retinal Layers) Measurements
Description: Using Spectral Domain optical coherence tomography (SD-OCT), horizontal macular thickness of the lamina cribrosa (boundaries of the retinal layers) is measured in the eyes of each participant in microohms.
Time Frame: 1 examination, approximately one hour
Measure: Mean (95% Confidence Interval); unit: micro-ohms
Groups:
- Open-angle Glaucoma Affected Eye: Affected eye of patients with primary open-angle glaucoma and visual field defect.
- Healthy Controls: Eyes of healthy controls with no glaucoma or other eye diseases.
- Open-angle Glaucoma Fellow Eye: Fellow eye of patients with primary open-angle glaucoma and no visual field defect.
Arm/Group | Open-angle Glaucoma Affected Eye | Healthy Controls | Open-angle Glaucoma Fellow Eye
Number analyzed (Participants) | 19 | 14 | 19
micro-ohms | 264.3 [258.3 to 270.3] | 273.3 [265.4 to 281.1] | 276.2 [270.0 to 282.4]

ADVERSE EVENTS:
Time Frame: 1 examination, approximately one hour
Groups:
- Open-angle Glaucoma: Participants with unilateral primary open-angle glaucoma (POAG) and visual field defect in only one eye.
- Healthy Controls: Participants without glaucoma and no other eye diseases.
Arm/Group | Open-angle Glaucoma | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14
Other Adverse Events (participants affected / at risk) | 0/19 | 0/14

LIMITATIONS AND CAVEATS:
Manual segmentation of macular layers, somewhat subjective measure, prone to errors of interpretation.

Cross sectional design did not allow for longitudinal tracking of fellow eyes. Pilot study was restricted by small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No